CLINICAL TRIAL: NCT00603382
Title: A Randomized Double-Blind, Double-Dummy, Placebo-Controlled, Parallel-Group, Multicenter, Dose Ranging Study to Evaluate the Efficacy and Safety of GW685698X Inhalation Powder Administered Once Daily and Fluticasone Propionate Inhalation Powder 100mcg Twice Daily Compared With Placebo for 8 Weeks in Adolescent and Adult Subjects With Persistent Asthma Symptomatic on Non-Steroidal, Asthma Therapy
Brief Title: A Randomized Study To Evaluate The Efficacy And Safety Of An Investigational Drug In Adolescent And Adult Subjects With Asthma Uncontrolled on Non-steroidal Therapy.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FFA109687
Record Dates: First submitted 2007-12-27; First posted 2008-01-29 (Estimated); Results first posted 2013-08-19 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-03

CONDITIONS: Asthma
Keywords: Adults; Pharmacokinetics; Pharmacogenetics; Asthma; Adolescents; GW685698X
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- GW685698X (Experimental)
  Interventions: Drug: GW685698X

INTERVENTIONS:
Drug: GW685698X — GW685698X
  Arms: GW685698X
Drug: Placebo — placebo comparator
  Arms: Placebo

SUMMARY:
This study is designed to determine if the investigational drug is effective and safe in individuals with asthma.

DETAILED DESCRIPTION:
A Randomized Double-Blind, Double-Dummy, Placebo-Controlled, Parallel-Group, Multicenter, Dose Ranging Study to Evaluate the Efficacy and Safety of GW685698X Inhalation Powder Once Daily and Fluticasone Propionate Inhalation Powder Twice Daily compared with Placebo for 8 Weeks in Adolescent and Adult Subjects with Persistent Asthma Symptomatic on Non-Steroidal, Asthma Therapy

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible for enrollment in the study must meet all of the following criteria:

* Type of Subject: Outpatient
* Age: 12 years of age or older at Visit 1. For sites in the following countries, subjects recruited will be ≥18 years of age: Bulgaria, Czech Republic, Germany, Greece, Lithuania, New Zealand, Russian Federation, Turkey and any other countries where local regulations or the regulatory status of study medication permit enrollment of adults only.
* Gender: Male or Eligible Female
* To be eligible for entry into the study, females of childbearing potential must commit to consistent and correct use of an acceptable method of birth control, as defined by the following:
* Male partner who is sterile prior to the female subject's entry into the study and is the sole sexual partner for that female subject
* Implants of levonorgestrel
* Injectable progestogen
* Oral contraceptive (either combined estrogen/progestin or progestin only)
* Any intrauterine device (IUD) with a documented failure rate of less than 1% per year.
* Females of childbearing potential who are not sexually active must commit to complete abstinence from intercourse throughout the clinical trial and for a period after the trial to account for elimination of the drug (minimum of six days).
* Double barrier method - spermicide plus a mechanical barrier (e.g., spermicide plus a male condom or a spermicide and female diaphragm).
* NB: For German sites, female subjects must use a method of birth control other than the double barrier method.
* The contraceptive transdermal patch, Ortho Evra (if the subject is less than 198 pounds)
* Female subjects should not be enrolled if they are pregnant, lactating or plan to become pregnant during the time of study participation. A serum pregnancy test is required of all females. This test will be performed at the initial screening visit (Visit 1) and Visit 8. In addition, a urine pregnancy test will be performed on the evening of the double-blind treatment visit, prior to randomization (Visit 3) and at Visits 4 through 7.
* Asthma Diagnosis: Asthma as defined by the National Institutes of Health [National Institutes of Health, 2007].
* Severity of Disease: A best FEV1 of 40%-85% of the predicted normal value during the morning Visit 1 screening period or a best FEV1 of 40%-90% of the predicted normal value during the evening Visit 1 screening period.
* Reversibility of Disease: Demonstrated a ≥ 12% and ≥200mL reversibility of FEV1 within approximately 30-minutes following 4 inhalations of albuterol/salbutamol inhalation aerosol (spacers are permitted for reversibility testing if required) or one nebulized albuterol/salbutamol solution at the screening period. Re-screening of subjects during the Visit 1 screening period: If a subject does not meet the inclusion criteria based upon FEV1 percent predicted and/or reversibility, the subject may return to the site once within 4 days and repeat the lung function tests.
* Current Anti-Asthma Therapy: Subjects must have been using a non-corticosteroid controller or short acting beta2-agonist bronchodilators alone (with no inhaled corticosteroids use for at least 6 weeks) for ≥ 3 months preceding Visit 1.
* Short- Acting Beta2-Agonists: All subjects must be able to replace their current short-acting beta2-agonists with albuterol/salbutamol inhalation aerosol at Visit 1 for use as needed for the duration of the study. The use of spacer devices with metered dose inhaler (MDI) or nebulized albuterol/salbutamol will not be allowed during the study with the exception of their use during reversibility testing at Visit 1. Subjects must be able to withhold all inhaled short-acting beta sympathomimetic bronchodilators for at least 6 hours prior to all study visits.
* Informed Consent: All subjects must be able and willing to give written informed consent to take part in the study.
* Compliance: Subjects must be able to comply with completion of the Daily Diary (includes paper medical conditions diary).
* French subjects: In France, a subject will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category.

Inclusion Criteria for Randomization

At the end of the run-in period, a subject will be eligible to enter the treatment period of the study if he/she meets the following criteria at Visit 3:

* Evening pre-dose percent predicted FEV1 of between 40% and 90% of their predicted normal.
* Any combination of the daily asthma symptom scores (day-time plus night-time) of ≥1 or albuterol/salbutamol use on at least 4 of the last 7 consecutive days of the run-in period (immediately preceding Visit 3).

Exclusion Criteria:

* History of Life-threatening asthma: Defined for this protocol as an asthma episode that required intubation and/or was associated with hypercapnia, respiratory arrest or hypoxic seizures.
* Respiratory Infection: Culture-documented or suspected bacterial or viral infection of the upper or lower respiratory tract, sinus or middle ear that is not resolved within 4 weeks before Visit 1 and led to a change in asthma management, or in the opinion of the Investigator is expected to affect the subjects asthma status or the subjects ability to participate in the study.
* Asthma Exacerbation: Any asthma exacerbation requiring oral corticosteroids within 3 months of Visit 1. A subject must not have had any hospitalization for asthma within 6 months prior to Visit 1.
* Concurrent Diseases/Abnormalities: Historical or current evidence of clinically significant uncontrolled disease including, but not limited to: cardiovascular disease, hepatic disease, renal disease, hematological disease, neurological disease, or pulmonary disease (including, but not confined to chronic bronchitis, emphysema, bronchiectasis with the need of treatment, cystic fibrosis, bronchopulmonary dysplasia, and chronic obstructive pulmonary disease). Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the subject at risk through participation, or which would affect the efficacy or safety analysis if the disease/condition exacerbated during the study. The list of additional excluded conditions/diseases includes, but is not limited to the following: congestive heart failure, clinically significant coronary heart disease, stroke within 3 months of Visit 1, poorly controlled peptic ulcer, immunologic compromise, tuberculosis (current or untreated), Addison's disease, uncontrolled thyroid disorder, known aortic aneurysm, clinically significant cardiac arrhythmia, uncontrolled hypertension1, hematological, hepatic, or renal disease, current malignancy2, cushings disease, uncontrolled diabetes mellitus, recent history of drug or alcohol abuse.
* systolic blood pressure ≥160, or diastolic blood pressure >100
* history of malignancy is acceptable only if subject has been in remission for one year prior to Visit 1 (remission = no current evidence of malignancy and no treatment for the malignancy in the 12 months prior to Visit 1)
* Patients with a history of tuberculosis who have received an approved prophylactic treatment regimen or an approved active treatment regimen and who have had no evidence of active disease for a minimum of 2 years may be enrolled [American Thoracic Society, 2003; American Thoracic Society, 2005]"
* Oropharyngeal Examination: A subject will not be eligible for the run-in if he/she has clinical visual evidence of oral candidiasis at Visit 1.
* Investigational Medications: A subject must not have participated in a study or used any investigational drug within 30 days prior to Visit 1.
* Drug Allergy: Any adverse reaction including immediate or delayed hypersensitivity to any beta2-agonist, sympathomimetic drug, or any intranasal, inhaled, or systemic corticosteroid therapy. Known or suspected sensitivity to the constituents of the novel dry powder inhaler or DISKUS/ACCUHALER (i.e., lactose or magnesium stearate).
* Milk Protein Allergy: History of severe milk protein allergy.
* Immunosuppressive Medications: A subject must not be using, or require use, of immunosuppressive medications during the study.

NOTE: Immunotherapy for the treatment of allergies is allowed during the study provided that the treatment was initiated prior to Visit 1 and the subject is maintained on a stable regimen throughout the study period.

* Attendance: A subject will not be eligible if he/she or his/her parent or legal guardian has any infirmity, disability, or geographical location which seems likely (in the opinion of the Investigator) to impair compliance with any aspect of this study protocol or scheduled visits to the study center and non-compliant with study medication or procedures (e.g. completion of daily diary). Neurological or psychiatric disease or history of drug or alcohol abuse which in the opinion of the investigator could interfere with the subject's proper completion of the protocol requirements excludes study participation.
* Tobacco Use : Current smoker or a smoking history of 10 pack years or more (e.g. 20 cigarettes/day for 10 years). A subject may not have used tobacco products within the past one year (i.e., cigarettes, cigars, or pipe tobacco).
* Affiliation with Investigator's Site: A subject will not be eligible for this study if he/she is an immediate family member of the participating Investigator, sub-Investigator, study coordinator, or employee of the participating Investigator.
* Corticosteroid Use: Administration of systemic, oral or depot corticosteroids within 12 weeks of Visit 1.

Administration of inhaled corticosteroids within 6 weeks of Visit 1.

* Potent Cytochrome P450 3A4 (CYP3A4) inhibitors: Patients who are receiving potent CYP3A4 inhibitors within 4 weeks of Visit 1 (e.g., ritonavir, ketoconazole, itraconazole).

Exclusion Criteria for Randomization At the end of the run-in period, a subject will not be eligible to enter the treatment period of the study if they meet any of the following criteria.

* Clinical Laboratory Abnormalities: Clinically significant abnormal laboratory tests during Visit 1 which are still abnormal upon repeat analysis and are not believed to be due to disease(s) present. Each Investigator will use his/her own discretion in determining the clinical significance of the abnormality. When in doubt, GlaxoSmithKline, or designee, should be notified so that a joint decision can be made.
* Changes in asthma medication (excluding albuterol/salbutamol inhalation aerosol provided at Visit 1).
* Occurrence of an culture-documented or suspected bacterial or viral infection of the upper or lower respiratory tract, sinus or middle ear during the run-in period that led to a change in asthma management, or in the opinion of the Investigator is expected to affect the subject's asthma status or the subject's ability to participate in the study.
* Asthma exacerbation, defined as any worsening of asthma requiring any treatment other than rescue albuterol/salbutamol or regular inhaled corticosteroid use. This includes requiring the use of systemic corticosteroids and / or emergency room visit or hospitalization or a change in subject's regular inhaled corticosteroid dose.
* A subject will not be eligible for randomization if he/she has an abnormal visual oropharyngeal exam at the randomization Visit 3 (visual clinical evidence of oral candidiasis).
* Non-compliance with completion of the Daily Diary, defined as: - Completion of AM and PM symptom scores on less than 4 days out of the last 7 days immediately preceding Visit 3.
* Completion of AM and PM rescue use on less than 4 days out of the last 7 days immediately preceding Visit 3.
* Completion of AM and PM PEF measurements on less than 4 days out of the last 7 days immediately preceding Visit 3.
* Recording run-in asthma medication use on less than 4 days out of the last 7 days immediately preceding Visit 3.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 599 (Actual)
Dates: Start 2007-12-01; Primary Completion 2008-10-01 (Actual); Study Completion 2008-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (135):
- United States (84):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Fort Smith, Arkansas
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Granada Hills, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Palmdale, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Roseville, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, West Covina, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Wheat Ridge, Colorado
  - GSK Investigational Site, Bridgeport, Connecticut
  - GSK Investigational Site, Waterbury, Connecticut
  - GSK Investigational Site, Boca Raton, Florida
  - GSK Investigational Site, Cocoa, Florida
  - GSK Investigational Site, Daytona Beach, Florida
  - GSK Investigational Site, Largo, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Winter Park, Florida
  - GSK Investigational Site, Gainesville, Georgia
  - GSK Investigational Site, Bloomingdale, Illinois
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, DeKalb, Illinois
  - GSK Investigational Site, Gurnee, Illinois
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Lenexa, Kansas
  - GSK Investigational Site, Crescent Springs, Kentucky
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Bangor, Maine
  - GSK Investigational Site, North Dartmouth, Massachusetts
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Taylor, Michigan
  - GSK Investigational Site, Ypsilanti, Michigan
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, Jackson, Mississippi
  - GSK Investigational Site, Rolla, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Warrensburg, Missouri
  - GSK Investigational Site, Billings, Montana
  - GSK Investigational Site, Butte, Montana
  - GSK Investigational Site, Missoula, Montana
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Clifton, New Jersey
  - GSK Investigational Site, Hillsborough, New Jersey
  - GSK Investigational Site, Red Bank, New Jersey
  - GSK Investigational Site, Skillman, New Jersey
  - GSK Investigational Site, East Syracuse, New York
  - GSK Investigational Site, Ithaca, New York
  - GSK Investigational Site, Rockville Centre, New York
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Greenville, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Eugene, Oregon
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Bluffton, South Carolina
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Boerne, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Dickinson, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Plano, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Waco, Texas
  - GSK Investigational Site, South Burlington, Vermont
  - GSK Investigational Site, Manassas, Virginia
  - GSK Investigational Site, Bellingham, Washington
  - GSK Investigational Site, Spokane, Washington
- Bulgaria (3):
  - GSK Investigational Site, Plovdiv
  - GSK Investigational Site, Sofia
  - GSK Investigational Site, Varna
- Canada (11):
  - GSK Investigational Site, Bay Roberts, Newfoundland and Labrador
  - GSK Investigational Site, Ajax, Ontario
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Mississauga, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Sainte-Foy, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
  - GSK Investigational Site, Trois-Rivières, Quebec
  - GSK Investigational Site, Saskatoon, Saskatchewan
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- France (6):
  - GSK Investigational Site, Évreux
  - GSK Investigational Site, Montbrison
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Toulon
  - GSK Investigational Site, Toulouse
  - GSK Investigational Site, Vieux-Condé
- Germany (5):
  - GSK Investigational Site, Sinsheim, Baden-Wurttemberg
  - GSK Investigational Site, Potsdam, Brandenburg
  - GSK Investigational Site, Gelnhausen, Hesse
  - GSK Investigational Site, Marburg, Hesse
  - GSK Investigational Site, Berlin
- Mexico (3):
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Zapopan, Jalisco
  - GSK Investigational Site, Monterrey N.L, Nuevo León
- GSK Investigational Site, Lima, Peru
- Philippines (3):
  - GSK Investigational Site, Cavite
  - GSK Investigational Site, Cebu City
  - GSK Investigational Site, Manila
- Poland (2):
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Zawadzkie
- Russia (5):
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Novokuznetsk
  - GSK Investigational Site, Samara
  - GSK Investigational Site, Smolensk
  - GSK Investigational Site, Yaroslavl
- Slovakia (3):
  - GSK Investigational Site, Banská Bystrica
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Martin
- South Korea (5):
  - GSK Investigational Site, Bucheon-si
  - GSK Investigational Site, Cheongju, Chungcheongbuk-do
  - GSK Investigational Site, Gwangju
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon, Kyonggi-do
- Sweden (2):
  - GSK Investigational Site, Boden
  - GSK Investigational Site, Luleå

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Bateman ED, Bleecker ER, Lotvall J, Woodcock A, Forth R, Medley H, Davis AM, Jacques L, Haumann B, Busse WW. Dose effect of once-daily fluticasone furoate in persistent asthma: a randomized trial. Respir Med. 2012 May;106(5):642-50. doi: 10.1016/j.rmed.2012.01.004. Epub 2012 Feb 18. PMID 22342538
- [Background] Psaila B, Bussel JB, Linden MD, Babula B, Li Y, Barnard MR, Tate C, Mathur K, Frelinger AL, Michelson AD. In vivo effects of eltrombopag on platelet function in immune thrombocytopenia: no evidence of platelet activation. Blood. 2012 Apr 26;119(17):4066-72. doi: 10.1182/blood-2011-11-393900. Epub 2012 Jan 31. PMID 22294727
- [Derived] O'Byrne PM, Jacques L, Goldfrad C, Kwon N, Perrio M, Yates LJ, Busse WW. Integrated safety and efficacy analysis of once-daily fluticasone furoate for the treatment of asthma. Respir Res. 2016 Nov 24;17(1):157. doi: 10.1186/s12931-016-0473-x. PMID 27881132
- [Derived] Gross AS, Goldfrad C, Hozawa S, James MH, Clifton CS, Sugiyama Y, Jacques L. Ethnic sensitivity assessment of fluticasone furoate/vilanterol in East Asian asthma patients from randomized double-blind multicentre Phase IIb/III trials. BMC Pulm Med. 2015 Dec 24;15:165. doi: 10.1186/s12890-015-0159-z. PMID 26704701
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: FFA109687 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: FFA109687 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: FFA109687 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: FFA109687 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: FFA109687 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: FFA109687 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: FFA109687 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants (par.) meeting eligibility criteria at the Screening visit completed a 28-day Run-in Period for Baseline, safety evaluations and measures of asthma status. Par. were then randomized to an 8-week Treatment Period. Total 1459 par. were screened, 601 were randomized of which 598 par. received at least one dose of study treatment.
Groups:
- Placebo: Participants received placebo once daily (OD) in the evening from the dry powder inhaler (DPI) and placebo twice daily (BID) from the DISKUS/ACCUHALER (one inhalation in the morning and one inhalation in the evening) for 8 weeks. In addition, participants were provided supplemental albuterol/salbutamol inhalation aerosol to be used as needed throughout the study.
- GW685698X 25 µg OD: Participants received GW685698X 25 micrograms (µg) OD in the evening from the DPI and placebo BID from the DISKUS/ACCUHALER (one inhalation in the morning and one inhalation in the evening) for 8 weeks. In addition, participants were provided supplemental albuterol/salbutamol aerosol to be used as needed throughout the study.
- GW685698X 50 µg OD: Participants received GW685698X 50 µg OD in the evening from the DPI and placebo BID from the DISKUS/ACCUHALER (one inhalation in the morning and one inhalation in the evening) for 8 weeks. In addition, participants were provided supplemental albuterol/salbutamol aerosol to be used as needed throughout the study.
- GW685698X 100 µg OD: Participants received GW685698X 100 µg OD in the evening from the DPI and placebo BID from the DISKUS/ACCUHALER (one inhalation in the morning and one inhalation in the evening) for 8 weeks. In addition, participants were provided supplemental albuterol/salbutamol aerosol to be used as needed throughout the study.
- GW685698X 200 µg OD: Participants received GW685698X 200 µg OD in the evening from the DPI and placebo BID from the DISKUS/ACCUHALER (one inhalation in the morning and one inhalation in the evening) for 8 weeks. In addition, participants were provided supplemental albuterol/salbutamol aerosol to be used as needed throughout the study.
- FP 100 µg BID: Participants received fluticasone propionate (FP) 100 µg BID from the DISKUS/ACCUHALER (one inhalation in the morning and one inhalation in the evening) plus placebo OD in the evening from the DPI for 8 weeks. In addition, participants were provided supplemental albuterol/salbutamol aerosol to be used as needed throughout the study.
Period: Overall Study
Arm/Group | Placebo | GW685698X 25 µg OD | GW685698X 50 µg OD | GW685698X 100 µg OD | GW685698X 200 µg OD | FP 100 µg BID
Started | 94 | 97 | 100 | 110 | 95 | 102
Completed | 76 | 83 | 91 | 98 | 86 | 84
Not Completed | 18 | 14 | 9 | 12 | 9 | 18
Not completed — Adverse Event | 0 | 1 | 1 | 2 | 1 | 2
Not completed — Lack of Efficacy | 14 | 9 | 3 | 6 | 6 | 11
Not completed — Protocol Violation | 1 | 0 | 1 | 2 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 1 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 2 | 0 | 1 | 3
Not completed — Withdrawal by Subject | 3 | 3 | 1 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants received placebo OD in the evening from the DPI and placebo BID from the DISKUS/ACCUHALER (one inhalation in the morning and one inhalation in the evening) for 8 weeks. In addition, participants were provided supplemental albuterol/salbutamol inhalation aerosol to be used as needed throughout the study.
- GW685698X 25 µg OD: Participants received GW685698X 25 µg OD in the evening from the DPI and placebo BID from the DISKUS/ACCUHALER (one inhalation in the morning and one inhalation in the evening) for 8 weeks. In addition, participants were provided supplemental albuterol/salbutamol aerosol to be used as needed throughout the study.
- FP 100 µg BID: Participants received FP 100 µg BID from the DISKUS/ACCUHALER (one inhalation in the morning and one inhalation in the evening) plus placebo OD in the evening from the DPI for 8 weeks. In addition, participants were provided supplemental albuterol/salbutamol aerosol to be used as needed throughout the study.
- Total: Total of all reporting groups
Arm/Group | Placebo | GW685698X 25 µg OD | GW685698X 50 µg OD | GW685698X 100 µg OD | GW685698X 200 µg OD | FP 100 µg BID | Total
Number analyzed (Participants) | 94 | 97 | 100 | 110 | 95 | 102 | 598
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.2 (15.82) | 37.7 (15.40) | 38.3 (14.49) | 36.8 (15.56) | 40.7 (15.96) | 39.9 (15.03) | 38.7 (15.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 57 | 59 | 60 | 60 | 56 | 339
  Male | 47 | 40 | 41 | 50 | 35 | 46 | 259
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African Heritage (AA/AHER) | 5 | 4 | 4 | 8 | 6 | 5 | 32
  American Indian or Alaska Native | 5 | 7 | 5 | 6 | 6 | 5 | 34
  Asian | 7 | 13 | 9 | 10 | 10 | 10 | 59
  White | 69 | 64 | 72 | 76 | 64 | 74 | 419
  AA/AHER & American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 1
  American Indian or Alaska Native & White | 8 | 8 | 9 | 10 | 8 | 8 | 51
  Native Hawaiian or other Pacific Islander & White | 0 | 1 | 1 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Trough (Evening Pre-dose and Pre- Rescue Bronchodilator) FEV1 at Week 8
Description: Pulmonary function was measured by forced expiratory volume in one second (FEV1), defined as the maximal amount of air that can be forcefully exhaled from the lungs in one second. Pre-dose and pre-rescue bronchodilator (albuterol/salbutamol) trough FEV1(the measurement of FEV1 performed at the end of the dosing interval) was measured electronically by spirometry in the evening at the Baseline through Week 8 clinic visits. Trough FEV1 is the FEV1 measured approximately 24 hours after the last administration of study drug. The highest of 3 technically acceptable measurements was recorded. The Visit 3 FEV1 assessment was used as the Baseline value. Change from Baseline in trough FEV1 was calculated as the value at Week 8 minus the value at Baseline. The analysis was performed using an Analysis of Covariance (ANCOVA) model with covariates of Baseline trough FEV1, country, sex, age, and treatment group.
Time Frame: Baseline and Week 8
Population: Intent-to-Treat (ITT) Population: all participants randomized to treatment who received at least one dose of study medication. The last observation carried forward (LOCF) method was used to impute missing data, in which the last non-missing post-BL on-treatment measurement (scheduled and unscheduled visits) was used to impute missing measurements.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | GW685698X 25 µg OD | GW685698X 50 µg OD | GW685698X 100 µg OD | GW685698X 200 µg OD | FP 100 µg BID
Number analyzed (Participants) | 93 | 94 | 97 | 109 | 94 | 101
Liters | 0.137 (0.0428) | 0.239 (0.0428) | 0.266 (0.0420) | 0.341 (0.0396) | 0.367 (0.0428) | 0.243 (0.0411)
Statistical Analysis 1: Comparison: Placebo vs GW685698X 25 µg OD; Test type: Superiority or Other; p = 0.095, ANCOVA; Median Difference (Final Values) = 0.101, 95% CI 2-sided [-0.018 to 0.221]
Statistical Analysis 2: Comparison: Placebo vs GW685698X 50 µg OD; Test type: Superiority or Other; p = 0.033, ANCOVA; Mean Difference (Final Values) = 0.129, 95% CI 2-sided [0.011 to 0.247]
Statistical Analysis 3: Comparison: Placebo vs GW685698X 100 µg OD; Test type: Superiority or Other; p < 0.001, ANCOVA; Median Difference (Final Values) = 0.204, 95% CI 2-sided [0.089 to 0.319]
Statistical Analysis 4: Comparison: Placebo vs GW685698X 200 µg OD; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.230, 95% CI 2-sided [0.111 to 0.349]
Statistical Analysis 5: Comparison: Placebo vs FP 100 µg BID; Test type: Superiority or Other; p = 0.074, ANCOVA; Mean Difference (Final Values) = 0.106, 95% CI 2-sided [-0.010 to 0.223]

2. Secondary Outcome: Mean Change From Baseline in Daily Trough (Pre-dose and Pre-rescue Bronchodilator) Evening Peak Expiratory Flow (PEF) Averaged Over the 8-week Treatment Period
Description: PEF is defined as the maximum airflow during a forced expiration beginning with the lungs fully inflated. Trough PEF is defined as the PEF measurement performed at the end of the dosing interval. PEF was measured by the participants using a hand-held electronic peak flow meter each evening prior to the dose of study medication and any rescue albuterol/salbutamol inhalation aerosol use. The best of three attempts was recorded by the participants in a daily diary. The Baseline value was derived from the last 7 days of the daily diary prior to the randomization of the participant. Change from Baseline was calculated as the value of the averaged daily evening PEF over the 8-week treatment period minus the value at Baseline. The analysis was performed using an ANCOVA model with covariates of Baseline trough evening PEF, country, sex, age, and treatment group.
Time Frame: From Baseline up to Week 8
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters per minute
Arm/Group | Placebo | GW685698X 25 µg OD | GW685698X 50 µg OD | GW685698X 100 µg OD | GW685698X 200 µg OD | FP 100 µg BID
Number analyzed (Participants) | 94 | 96 | 98 | 110 | 95 | 102
Liters per minute | 9.6 (4.21) | 23.6 (4.17) | 30.3 (4.12) | 25.7 (3.90) | 31.3 (4.20) | 24.4 (4.04)

3. Secondary Outcome: Mean Change From Baseline in Daily Morning PEF Averaged Over the 8-week Treatment Period
Description: PEF is defined as the maximum airflow during a forced expiration beginning with the lungs fully inflated. Trough PEF is defined as the PEF measurement performed at th end of the dosing interval. PEF was measured by the participants using a hand-held electronic peak flow meter each morning prior to the dose of study medication and any rescue albuterol/salbutamol inhalation aerosol use. The best of three attempts was recorded by the participants in a daily diary. The Baseline value was derived from the last 7 days of the daily diary prior to the randomization of the participant. Change from Baseline was calculated as the value of the averaged daily morning PEF over the 8-week treatment period minus the value at Baseline. The analysis was performed using an ANCOVA model with covariates of Baseline trough morning PEF, country, sex, age, and treatment group.
Time Frame: From Baseline up to Week 8
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters per minute
Arm/Group | Placebo | GW685698X 25 µg OD | GW685698X 50 µg OD | GW685698X 100 µg OD | GW685698X 200 µg OD | FP 100 µg BID
Number analyzed (Participants) | 94 | 96 | 98 | 110 | 95 | 102
Liters per minute | 13.6 (4.27) | 27.2 (4.23) | 33.5 (4.17) | 29.5 (3.95) | 35.6 (4.26) | 25.6 (4.09)

4. Secondary Outcome: Mean Change From Baseline in the Percentage of Symptom-free 24 Hour (hr) Periods During the 8-week Treatment Period
Description: Asthma symptoms were recorded in a daily dairy by the participants every day in the morning and evening before taking any rescue or study medication and before PEF measurement. A 24-hour period in which a participant's responses to both the morning and evening assessments indicated no symptoms was considered as symptom-free. The Baseline value was derived from the last 7 days of the daily diary prior to the randomization of the participant. Change from Baseline was calculated as the averaged value during the 8-week Treatment Period minus the value at Baseline. The analysis was performed using an ANCOVA model with covariates of Baseline, country, sex, age, and treatment group.
Time Frame: From Baseline up to Week 8
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of symptom-free 24-hr periods
Arm/Group | Placebo | GW685698X 25 µg OD | GW685698X 50 µg OD | GW685698X 100 µg OD | GW685698X 200 µg OD | FP 100 µg BID
Number analyzed (Participants) | 94 | 96 | 98 | 110 | 95 | 102
Percentage of symptom-free 24-hr periods | 18.4 (3.21) | 25.3 (3.17) | 31.1 (3.14) | 38.7 (2.97) | 31.7 (3.20) | 33.3 (3.08)

5. Secondary Outcome: Mean Change From Baseline in the Percentage of Rescue Free 24-hour (hr) Periods During the 8-week Treatment Period
Description: The number of inhalations of rescue albuterol/salbutamol inhalation aerosol used during the day and night was recorded by the participants in a daily diary. A 24-hour period in which a participant's responses to both the morning and evening assessments indicated no use of rescue medication was considered as rescue-free. The Baseline value was derived from the last 7 days of the daily diary prior to the randomization of the participant. Change from Baseline was calculated as the averaged value during the 8-week Treatment Period minus the value at Baseline. The analysis was performed using an ANCOVA model with covariates of Baseline, country, sex, age, and treatment group.
Time Frame: From Baseline up to Week 8
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of rescue-free 24-hr periods
Arm/Group | Placebo | GW685698X 25 µg OD | GW685698X 50 µg OD | GW685698X 100 µg OD | GW685698X 200 µg OD | FP 100 µg BID
Number analyzed (Participants) | 94 | 96 | 98 | 110 | 95 | 102
Percentage of rescue-free 24-hr periods | 21.9 (3.32) | 29.3 (3.28) | 34.5 (3.24) | 40.8 (3.08) | 32.0 (3.31) | 35.5 (3.18)

6. Secondary Outcome: Number of Participants Who Withdrew Due to Lack of Efficacy During the 8-Week Treatment Period
Description: The number of participants whose primary reason for withdrawal was lack of efficacy was analyzed.
Time Frame: From the first dose of study medication up to Week 8/Early Withdrawal
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo | GW685698X 25 µg OD | GW685698X 50 µg OD | GW685698X 100 µg OD | GW685698X 200 µg OD | FP 100 µg BID
Number analyzed (Participants) | 94 | 97 | 100 | 110 | 95 | 102
participants | 14 | 9 | 3 | 6 | 6 | 11

7. Secondary Outcome: Number of Participants With Any On-treatment Adverse Events or Serious Adverse Events Throughout the 8-week Treatment Period
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A serious adverse event (SAE) is defined as any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires hospitalization or prolongation of existing hospitalization; results in disability/incapacity; or is a congenital anomaly/birth defect. Medical or scientific judgment should have been exercised in other situations. Refer to the general AE/SAE module for a list of AEs (occurring at a frequency threshold >=3%) and SAEs.
Time Frame: From the first dose of study medication up to Week 8/Early Withdrawal
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo | GW685698X 25 µg OD | GW685698X 50 µg OD | GW685698X 100 µg OD | GW685698X 200 µg OD | FP 100 µg BID
Number analyzed (Participants) | 94 | 97 | 100 | 110 | 95 | 102
participants
  Any AE | 24 | 19 | 28 | 35 | 27 | 35
  Any SAE | 0 | 1 | 0 | 1 | 0 | 2

8. Secondary Outcome: Number of Participants With Clinical/Visual Evidence of Oropharyngeal Candidiasis
Description: A detailed oropharyngeal examination for visual evidence of oral candidiasis was performed.
Time Frame: From Baseline up to Week 8/Early Withdrawal
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo | GW685698X 25 µg OD | GW685698X 50 µg OD | GW685698X 100 µg OD | GW685698X 200 µg OD | FP 100 µg BID
Number analyzed (Participants) | 94 | 97 | 100 | 110 | 95 | 102
participants
  Clinical evidence | 0 | 0 | 4 | 4 | 2 | 2
  No clinical evidence | 94 | 97 | 96 | 106 | 93 | 100

9. Secondary Outcome: Percentage of Basophils, Eosinophils, Lymphocytes, Monocytes, and Total Neutrophils in the Blood at Baseline and Week 8
Description: Blood samples were collected for the measurement of basophils, eosinophils, lymphocytes, monocytes, and total neutrophils at Baseline (BL) and Week 8 (W8). The Baseline value was the measurement taken at screening (Visit 1).
Time Frame: Baseline and Week 8
Population: ITT Population. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles). Different participants may have been analyzed for different parameters, so the overall number of participants analyzed reflects everyone in the ITT Population.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Placebo | GW685698X 25 µg OD | GW685698X 50 µg OD | GW685698X 100 µg OD | GW685698X 200 µg OD | FP 100 µg BID
Number analyzed (Participants) | 94 | 97 | 100 | 110 | 95 | 102
Percentage
  Basophils, BL, n=92, 94, 95, 106, 92, 97 | 0.31 (0.199) | 0.32 (0.200) | 0.31 (0.194) | 0.32 (0.190) | 0.33 (0.205) | 0.33 (0.234)
  Basophils,W8, n=72, 80, 83, 94, 82, 79 | 0.30 (0.186) | 0.26 (0.153) | 0.31 (0.169) | 0.35 (0.236) | 0.35 (0.220) | 0.34 (0.264)
  Eosinophils, BL, n=92, 94, 95, 106, 92, 97 | 3.87 (3.022) | 3.38 (2.693) | 3.95 (2.503) | 4.40 (3.286) | 4.75 (3.358) | 3.88 (3.073)
  Eosinophils, W8, n=72, 80, 83, 94, 82, 79 | 4.31 (3.544) | 3.38 (3.300) | 3.76 (2.608) | 3.77 (3.066) | 3.96 (2.867) | 3.34 (2.364)
  Lymphocytes, BL, n=92, 94, 95, 106, 92, 97 | 33.96 (8.378) | 31.57 (8.821) | 33.33 (7.768) | 33.69 (8.682) | 34.32 (8.806) | 34.25 (8.514)
  Lymphocytes, W8, n=72, 80, 83, 94, 82, 79 | 32.88 (8.063) | 29.82 (10.120) | 30.36 (8.322) | 30.39 (7.326) | 31.97 (7.440) | 32.22 (7.877)
  Monocytes, BL, n=92, 94, 95, 106, 92, 97 | 5.09 (2.379) | 4.41 (1.851) | 4.70 (2.056) | 5.20 (2.113) | 4.78 (2.301) | 4.92 (2.093)
  Monocytes, W8, n=72, 80, 83, 94, 82, 79 | 5.41 (3.042) | 4.32 (2.098) | 4.60 (2.486) | 4.60 (2.178) | 4.50 (2.174) | 4.87 (2.380)
  Total Neutrophils, BL, n=92, 94, 95, 106, 92, 97 | 56.74 (9.220) | 60.24 (9.620) | 57.68 (8.309) | 56.34 (9.832) | 55.80 (10.281) | 56.60 (9.226)
  Total Neutrophils, W8, n=72, 80, 83, 94, 82, 79 | 57.08 (9.543) | 62.19 (11.580) | 60.95 (9.008) | 60.86 (8.054) | 59.20 (8.881) | 59.19 (8.672)

10. Secondary Outcome: Hematocrit at Baseline and Week 8
Description: Blood samples were collected for the measurement of Hematocrit at Baseline (BL) and Week 8 (W8). The Baseline value was the measurement taken at screening (Visit 1).
Time Frame: Baseline and Week 8
Population: ITT Population. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the ITT Population.
Measure: Mean (Standard Deviation); unit: Proportion of 1
Arm/Group | Placebo | GW685698X 25 µg OD | GW685698X 50 µg OD | GW685698X 100 µg OD | GW685698X 200 µg OD | FP 100 µg BID
Number analyzed (Participants) | 94 | 97 | 100 | 110 | 95 | 102
Proportion of 1
  Hematocrit, BL, n=92, 94, 95, 106, 92, 97 | 0.43 (0.041) | 0.42 (0.039) | 0.42 (0.040) | 0.43 (0.043) | 0.42 (0.039) | 0.43 (0.034)
  Hematocrit, W8, n=72, 79, 83, 94, 82, 79 | 0.43 (0.038) | 0.42 (0.038) | 0.42 (0.037) | 0.43 (0.040) | 0.42 (0.033) | 0.43 (0.039)

11. Secondary Outcome: Hemoglobin at Baseline and Week 8
Description: Blood samples were collected for the measurement of hemoglobin at Baseline (BL)and Week 8 (W8). The Baseline value was the measurement taken at screening (Visit 1).
Time Frame: Baseline and Week 8
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Grams per liter (G/L)
Arm/Group | Placebo | GW685698X 25 µg OD | GW685698X 50 µg OD | GW685698X 100 µg OD | GW685698X 200 µg OD | FP 100 µg BID
Number analyzed (Participants) | 94 | 97 | 100 | 110 | 95 | 102
Grams per liter (G/L)
  Hemoglobin, BL, n=92, 94, 95, 106, 92, 96 | 141.54 (14.116) | 138.05 (13.178) | 140.70 (13.769) | 141.14 (14.625) | 139.50 (12.978) | 141.90 (11.632)
  Hemoglobin, W8, n=72, 79, 83, 94, 82, 79 | 140.81 (12.973) | 137.86 (12.862) | 138.95 (12.785) | 140.16 (13.647) | 136.32 (11.594) | 139.81 (13.009)

12. Secondary Outcome: Platelet Count and White Blood Cell (WBC) Count at Baseline and Week 8
Description: Blood samples were collected for the measurement of platelet count and WBC count at Baseline (BL) and Week 8 (W8). The Baseline value was the measurement taken at screening (Visit 1).
Time Frame: Baseline and Week 8
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter (GI/L)
Arm/Group | Placebo | GW685698X 25 µg OD | GW685698X 50 µg OD | GW685698X 100 µg OD | GW685698X 200 µg OD | FP 100 µg BID
Number analyzed (Participants) | 94 | 97 | 100 | 110 | 95 | 102
10^9 cells per liter (GI/L)
  Platelet count, BL, n=91, 91, 95, 106, 92, 95 | 271.68 (62.861) | 265.75 (51.446) | 279.38 (57.658) | 272.20 (61.111) | 268.37 (60.442) | 281.26 (66.492)
  Platelet count, W8, n=72, 76, 83, 93, 81, 78 | 265.47 (49.978) | 262.07 (45.837) | 271.03 (47.156) | 278.57 (58.302) | 272.53 (68.404) | 274.46 (61.819)
  WBC, BL, n=92, 94, 95, 106, 92, 97 | 7.82 (2.018) | 7.96 (1.892) | 8.01 (2.095) | 7.62 (1.878) | 7.79 (2.055) | 7.94 (1.982)
  WBC, W8, n=72, 79, 83, 94, 82, 79 | 7.56 (1.679) | 8.26 (2.169) | 8.34 (2.211) | 7.94 (2.046) | 7.94 (1.769) | 8.00 (2.292)

13. Secondary Outcome: Red Blood Cells (RBC) Count at Baseline and Week 8
Description: Blood samples were collected for the measurement of RBC count at Baseline (BL) and Week 8 (W8). The Baseline value was the measurement taken at screening (Visit 1).
Time Frame: Baseline and Week 8
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter (TI/L)
Arm/Group | Placebo | GW685698X 25 µg OD | GW685698X 50 µg OD | GW685698X 100 µg OD | GW685698X 200 µg OD | FP 100 µg BID
Number analyzed (Participants) | 94 | 97 | 100 | 110 | 95 | 102
10^12 cells per liter (TI/L)
  RBC, BL, n=92, 94, 95, 106, 92, 97 | 4.71 (0.429) | 4.65 (0.438) | 4.68 (0.425) | 4.71 (0.460) | 4.68 (0.422) | 4.71 (0.416)
  RBC, W8, n=72, 79, 83, 94, 82, 79 | 4.65 (0.410) | 4.61 (0.445) | 4.63 (0.435) | 4.67 (0.450) | 4.60 (0.369) | 4.65 (0.462)

14. Secondary Outcome: Clinical Chemistry Parameters of Alkaline Phosphatase (ALP), Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Lactate Dehydrogenase (LD), and Gamma Glutamyltransferase (GGT) at Baseline and Week 8
Description: Blood samples were collected for the measurement of ALP, ALT, AST, LD and GGT at Baseline (BL) and Week 8 (W8). The Baseline value was the measurement taken at Screening (Visit 1).
Time Frame: Baseline and Week 8
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | Placebo | GW685698X 25 µg OD | GW685698X 50 µg OD | GW685698X 100 µg OD | GW685698X 200 µg OD | FP 100 µg BID
Number analyzed (Participants) | 94 | 97 | 100 | 110 | 95 | 102
International units per liter (IU/L)
  ALP, BL, n=94, 97, 99, 106, 94, 101 | 82.7 (36.11) | 79.7 (32.21) | 83.5 (40.07) | 90.3 (56.43) | 94.4 (71.94) | 84.7 (62.31)
  ALP, W8, n=78, 84, 90, 97, 85, 83 | 83.0 (40.83) | 74.8 (27.91) | 82.9 (41.61) | 87.0 (49.65) | 90.8 (76.22) | 84.0 (59.81)
  ALT, BL, n=94, 97, 99, 106, 94, 101 | 21.8 (15.91) | 21.5 (14.57) | 23.6 (19.40) | 22.3 (16.61) | 20.7 (11.38) | 20.1 (9.84)
  ALT, W8, n=78, 84, 90, 97, 86, 83 | 22.3 (22.79) | 20.3 (11.92) | 20.7 (10.39) | 20.8 (14.01) | 19.5 (12.03) | 19.9 (10.04)
  AST, BL, n=94, 96, 99, 105, 93, 101 | 21.0 (7.64) | 22.8 (11.39) | 22.8 (13.35) | 21.9 (9.68) | 21.3 (7.20) | 20.3 (5.10)
  AST, W8, n=78, 83, 90, 97, 86, 82 | 22.2 (10.76) | 20.8 (6.48) | 21.1 (7.52) | 20.5 (8.07) | 20.2 (5.91) | 20.5 (5.38)
  LD, BL, n=94, 96, 99, 105, 93, 101 | 157.9 (47.78) | 170.7 (59.82) | 169.3 (64.08) | 165.6 (70.56) | 172.9 (62.38) | 164.2 (57.04)
  LD, W8, n=78, 83, 90, 97, 86, 82 | 151.8 (32.37) | 159.1 (31.46) | 159.9 (32.14) | 153.8 (26.90) | 161.9 (36.79) | 157.3 (27.36)
  GGT, BL, n=94, 97, 99, 106, 94, 101 | 27.6 (20.00) | 33.0 (30.67) | 33.1 (31.42) | 30.1 (22.29) | 29.9 (26.30) | 28.2 (21.40)
  GGT, W8, n=78, 84, 90, 97, 86, 83 | 29.7 (27.53) | 31.1 (24.61) | 32.4 (30.84) | 31.9 (24.96) | 29.3 (32.75) | 27.9 (21.24)

15. Secondary Outcome: Clinical Chemistry Parameters of Albumin and Total Protein at Baseline and Week 8
Description: Blood samples were collected for the measurement of albumin and total protein at Baseline (BL) and Week 8 (W8). The Baseline value was the measurement taken at Screening (Visit 1).
Time Frame: Baseline and Week 8
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | Placebo | GW685698X 25 µg OD | GW685698X 50 µg OD | GW685698X 100 µg OD | GW685698X 200 µg OD | FP 100 µg BID
Number analyzed (Participants) | 94 | 97 | 100 | 110 | 95 | 102
Grams per liter (g/L)
  Albumin,BL, n=94, 97, 99, 106, 94, 101 | 45.2 (3.18) | 45.6 (3.08) | 45.1 (2.86) | 45.9 (3.00) | 45.3 (2.96) | 45.2 (3.01)
  Albumin, W8, n= 78, 84, 90, 97, 86, 83 | 44.9 (3.12) | 44.8 (3.30) | 44.9 (2.97) | 45.6 (2.91) | 44.5 (3.22) | 44.9 (2.62)
  Total protein, BL, n=94, 97, 99, 106, 94, 101 | 73.2 (4.04) | 74.0 (4.46) | 73.1 (4.60) | 74.1 (4.63) | 73.4 (4.50) | 73.2 (4.23)
  Total protein, W8, n= 78, 84, 90, 97, 86, 83 | 71.9 (3.65) | 72.6 (4.21) | 72.6 (4.62) | 73.4 (4.58) | 72.0 (4.66) | 72.5 (4.05)

16. Secondary Outcome: Clinical Chemistry Parameters of Chloride, Calcium, Carbon Dioxide Content/Bicarbonate (CO2/BI), Cholesterol, Glucose, Phosphorus Inorganic(PI), Potassium, Sodium, and Urea/Blood Urea Nitrogen (BUN) at Baseline and Week 8
Description: Blood samples were collected for the measurement of chloride, calcium, CO2/BI, cholesterol, glucose, PI, potassium, sodium, and urea/blood urea nitrogen at Baseline (BL) and Week 8 (W8). The Baseline value was the measurement taken at screening (Visit 1).
Time Frame: Baseline and Week 8
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Placebo | GW685698X 25 µg OD | GW685698X 50 µg OD | GW685698X 100 µg OD | GW685698X 200 µg OD | FP 100 µg BID
Number analyzed (Participants) | 94 | 97 | 100 | 110 | 95 | 102
Millimoles per liter (mmol/L)
  Chloride, BL, n=94, 97, 99, 106, 94, 101 | 104.4 (2.25) | 104.7 (2.38) | 104.5 (2.50) | 104.4 (2.41) | 104.8 (2.17) | 104.4 (2.49)
  Chloride, W8, n=78, 84, 90, 97, 86, 83 | 104.8 (2.24) | 104.8 (2.36) | 104.7 (2.55) | 104.2 (2.15) | 104.7 (2.11) | 104.6 (2.67)
  Calcium, BL, n=94, 96, 99, 105, 93, 101 | 2.4 (0.10) | 2.4 (0.10) | 2.3 (0.09) | 2.4 (0.11) | 2.4 (0.13) | 2.3 (0.09)
  Calcium, W8, n=78, 83, 90, 97, 85, 82 | 2.4 (0.10) | 2.3 (0.10) | 2.3 (0.10) | 2.4 (0.10) | 2.4 (0.11) | 2.4 (0.09)
  CO2/BI, BL, n=94, 96, 99, 105, 93, 101 | 23.2 (2.58) | 22.8 (2.71) | 23.0 (2.31) | 23.4 (2.49) | 23.5 (2.45) | 23.5 (2.74)
  CO2/BI, W8, n=78, 83, 90, 97, 86, 82 | 23.1 (2.57) | 22.8 (2.62) | 22.7 (2.61) | 23.3 (2.55) | 22.7 (2.42) | 22.8 (2.60)
  Cholesterol, BL, n=94, 97, 99, 106, 94, 101 | 4.9 (1.02) | 5.0 (1.04) | 5.2 (1.14) | 5.0 (0.97) | 5.0 (1.08) | 5.0 (1.10)
  Cholesterol, W8, n=78, 84, 90, 97, 86, 83 | 5.0 (1.24) | 4.9 (1.05) | 5.1 (1.05) | 5.2 (1.16) | 5.0 (1.03) | 5.0 (1.07)
  Glucose, BL, n=94, 97, 99, 106, 94, 101 | 5.2 (0.99) | 5.5 (2.05) | 5.2 (1.18) | 5.1 (0.89) | 5.1 (0.83) | 5.3 (1.54)
  Glucose, W8, n=78, 84, 90, 97, 86, 83 | 5.2 (1.07) | 5.4 (1.96) | 5.2 (1.20) | 5.0 (0.88) | 5.2 (1.21) | 5.1 (1.18)
  PI, BL, n=94, 97, 99, 106, 94, 101 | 1.2 (0.22) | 1.1 (0.20) | 1.2 (0.17) | 1.2 (0.22) | 1.2 (0.21) | 1.2 (0.18)
  PI, W8, n=78, 84, 90, 97, 86, 83 | 1.3 (0.21) | 1.2 (0.17) | 1.2 (0.18) | 1.3 (0.20) | 1.2 (0.21) | 1.2 (0.20)
  Potassium, BL, n=94, 96, 99, 105, 93, 101 | 4.1 (0.39) | 4.2 (0.44) | 4.1 (0.38) | 4.2 (0.40) | 4.2 (0.45) | 4.2 (0.40)
  Potassium, W8, n=78, 83, 90, 97, 85, 82 | 4.2 (0.34) | 4.2 (0.41) | 4.2 (0.32) | 4.2 (0.38) | 4.2 (0.38) | 4.2 (0.36)
  Sodium, BL, n=94, 97, 99, 106, 94, 101 | 140.8 (1.82) | 140.5 (2.05) | 140.6 (1.92) | 140.8 (2.16) | 141.1 (1.91) | 140.8 (2.04)
  Sodium, W8, n=78, 84, 90, 97, 86, 83 | 140.7 (2.09) | 140.5 (2.01) | 140.7 (2.02) | 140.6 (1.63) | 140.9 (2.36) | 140.8 (1.97)
  BUN, BL, n=94, 97, 99, 106, 94, 101 | 5.4 (1.75) | 5.3 (1.66) | 5.3 (1.92) | 5.7 (1.94) | 5.7 (2.09) | 5.4 (1.72)
  BUN, W8, n=78, 84, 90, 97, 86, 83 | 5.5 (1.68) | 5.2 (1.97) | 5.0 (1.30) | 5.5 (1.44) | 5.2 (1.54) | 5.0 (1.43)

17. Secondary Outcome: Clinical Chemistry Parameters of Creatinine, Direct Bilirubin, Total Bilirubin, and Uric Acid at Baseline and Week 8
Description: Blood samples were collected for the measurement of creatinine, direct bilirubin (DBIL), total bilirubin (TBIL), and uric acid at Baseline and Week 8. The Baseline value was the measurement taken at screening (Visit 1).
Time Frame: Baseline and Week 8
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Micromoles per liter (µmol/L)
Arm/Group | Placebo | GW685698X 25 µg OD | GW685698X 50 µg OD | GW685698X 100 µg OD | GW685698X 200 µg OD | FP 100 µg BID
Number analyzed (Participants) | 94 | 97 | 100 | 110 | 95 | 102
Micromoles per liter (µmol/L)
  DBIL, BL, n=94, 97, 99, 106, 94, 101 | 2.1 (1.26) | 2.1 (1.29) | 2.0 (1.04) | 2.0 (1.13) | 1.8 (1.17) | 2.0 (1.04)
  DBIL, W8, n=77, 84, 89, 97, 86, 83 | 2.0 (1.03) | 2.0 (0.94) | 1.9 (0.98) | 1.9 (1.02) | 1.7 (0.93) | 1.9 (1.05)
  TBIL, BL, n=94, 97, 99, 106, 94, 101 | 9.6 (6.10) | 9.7 (6.08) | 9.0 (4.39) | 9.3 (4.35) | 8.7 (4.11) | 9.0 (3.93)
  TBIL, W8, n=78, 84, 90, 97, 86, 83 | 10.3 (5.57) | 9.1 (4.14) | 8.7 (3.99) | 9.1 (3.88) | 8.5 (3.46) | 9.4 (4.39)
  Uric acid, BL, n=94, 97, 99, 105, 94, 101 | 337.8 (88.15) | 327.2 (85.64) | 325.6 (85.82) | 334.1 (90.63) | 326.6 (85.37) | 324.5 (78.64)
  Uric acid, W8, n=78, 84, 90, 96, 86, 83 | 353.6 (86.64) | 327.5 (84.69) | 321.9 (91.90) | 340.9 (89.48) | 316.5 (81.29) | 325.4 (80.48)
  Creatinine, BL, n=94, 97, 99, 106, 94, 101 | 83.2 (19.89) | 79.8 (14.72) | 77.7 (14.52) | 81.9 (16.68) | 78.3 (15.21) | 79.3 (15.08)
  Creatinine, W8, n=78, 84, 90, 97, 86, 83 | 84.5 (19.21) | 79.7 (15.67) | 79.0 (13.45) | 81.7 (14.90) | 77.7 (14.32) | 80.4 (15.97)

18. Secondary Outcome: Number of Participants With the Indicated Result for the Indicated Urinalysis Parameters Tested by Dipstick at Baseline and Week 8/Early Withdrawal
Description: Urinalysis parameters included: Urine Occult Blood (UOB), Urine Glucose (UG), Urine Ketones (UK), Urine Protein (UP), and Urine Leukocyte Esterase test for detecting White Blood Cell (UWBC). The dipstick was a strip used to detect the presence or absence of these parameters in the urine sample. The dipstick test gives results in a semi-quantitative manner, and results for urinalysis parameters can be read as large, moderate (Mod), negative (Neg), small, Trace, 1+, 2+, 3+ and 4+, and for UG the result can be read as Neg, Trace, Trace or 1/10 G/dL, 1+ or 1/4 G/dL, 3+ or 1 G/dL, indicating proportional concentrations in the urine sample. Data are reported as the number of participants who had neg, Trace, 1+, 2+, 3+ and 4+ levels at Baseline (BL) and Week 8 (W8)/Early Withdrawal (EW). The Baseline value was the measurement taken at screening (Visit 1).
Time Frame: Baseline and Week 8/Early Withdrawal
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | Placebo | GW685698X 25 µg OD | GW685698X 50 µg OD | GW685698X 100 µg OD | GW685698X 200 µg OD | FP 100 µg BID
Number analyzed (Participants) | 94 | 97 | 100 | 110 | 95 | 102
participants
  UOB, 1+, BL, n=92, 94, 95, 106, 93, 96 | 2 | 1 | 3 | 4 | 3 | 2
  UOB, 2+, BL, n=92, 94, 95, 106, 93, 96 | 3 | 1 | 2 | 0 | 1 | 1
  UOB, 3+, BL, n=92, 94, 95, 106, 93, 96 | 2 | 0 | 0 | 2 | 2 | 2
  UOB, 4+, BL, n=92, 94, 95, 106, 93, 96 | 0 | 0 | 0 | 1 | 0 | 0
  UOB, Mod, BL, n=92, 94, 95, 106, 93, 96 | 1 | 0 | 0 | 0 | 0 | 1
  UOB, Neg, BL, n=92, 94, 95, 106, 93, 96 | 79 | 91 | 83 | 97 | 81 | 82
  UOB, Small, BL, n=92, 94, 95, 106, 93, 96 | 0 | 0 | 3 | 0 | 1 | 0
  UOB, Trace, BL, n=92, 94, 95, 106, 93, 96 | 5 | 1 | 4 | 2 | 5 | 8
  UOB, 1+, W8, n=71, 81, 82, 93, 82, 77 | 1 | 1 | 1 | 0 | 4 | 3
  UOB, 2+, W8, n=71, 81, 82, 93, 82, 77 | 4 | 2 | 2 | 2 | 2 | 3
  UOB, 3+, W8, n=71, 81, 82, 93, 82, 77 | 0 | 3 | 0 | 0 | 0 | 1
  UOB, Large, W8, n=71, 81, 82, 93, 82, 77 | 0 | 0 | 0 | 0 | 1 | 0
  UOB, Mod, W8, n=71, 81, 82, 93, 82, 77 | 0 | 0 | 0 | 0 | 1 | 0
  UOB, Neg, W8, n=71, 81, 82, 93, 82, 77 | 62 | 71 | 73 | 83 | 69 | 66
  UOB, Trace, W8, n=71, 81, 82, 93, 82, 77 | 4 | 4 | 6 | 8 | 5 | 4
  UOB, Neg, EW, n=2, 1, 2, 3, 1, 7 | 2 | 1 | 2 | 3 | 1 | 7
  UG, 1+ or 1/4 G/DL, BL, n=92, 94, 95, 106, 93, 96 | 0 | 0 | 0 | 0 | 0 | 1
  UG, 3+ or 1 G/DL, BL, n=92, 94, 95, 106, 93, 96 | 0 | 2 | 1 | 0 | 0 | 1
  UG, 4+ or 2 or more G/DL, n=92, 94, 95, 106, 93,96 | 0 | 1 | 0 | 0 | 0 | 0
  UG, Neg, BL, n=92, 94, 95, 106, 93, 96 | 90 | 91 | 94 | 105 | 91 | 94
  UG, Trace, BL, n=92, 94, 95, 106, 93, 96 | 1 | 0 | 0 | 1 | 1 | 0
  UG, Trace or 1/10 G/DL, BL, n=92, 94, 95,106,93,96 | 1 | 0 | 0 | 0 | 1 | 0
  UG, 1+ or 1/4 G/DL, W8, n=71, 81, 82, 93, 82, 77 | 0 | 1 | 1 | 0 | 0 | 0
  UG, 3+ or 1 G/DL, W8, n=71, 81, 82, 93, 82, 77 | 0 | 3 | 1 | 0 | 0 | 1
  UG, Neg, W8, n=71, 81, 82, 93, 82, 77 | 71 | 77 | 80 | 92 | 78 | 76
  UG, Trace, W8, n=71, 81, 82, 93, 82, 77 | 0 | 0 | 0 | 0 | 2 | 0
  UG, Trace or 1/10 G/DL, W8, n=71, 81, 82, 93,82,77 | 0 | 0 | 0 | 1 | 2 | 0
  UG, Neg, EW, n=2, 1, 2, 3, 1, 7 | 2 | 1 | 2 | 3 | 1 | 7
  UK, 1+, BL, n=92, 94, 95, 106, 93, 96 | 0 | 0 | 1 | 1 | 1 | 0
  UK, 2+, BL, n=92, 94, 95, 106, 93, 96 | 0 | 0 | 0 | 0 | 1 | 0
  UK, Neg, BL, n=92, 94, 95, 106, 93, 96 | 91 | 89 | 92 | 104 | 90 | 95
  UK, Trace, BL, n=92, 94, 95, 106, 93, 96 | 1 | 5 | 2 | 1 | 1 | 1
  UK, 2+, W8, n=71, 81, 82, 93, 82, 77 | 0 | 0 | 0 | 1 | 0 | 0
  UK, Neg, W8, n=71, 81, 82, 93, 82, 77 | 67 | 77 | 78 | 91 | 79 | 69
  UK, Trace, W8, n=71, 81, 82, 93, 82, 77 | 4 | 4 | 4 | 1 | 3 | 8
  UK, Neg, EW, n=2, 1, 2, 3, 1, 7 | 2 | 1 | 2 | 3 | 1 | 7
  UP, 1+, BL, n=92, 94, 95, 106, 93, 96 | 7 | 7 | 6 | 8 | 5 | 4
  UP, 2+, BL, n=92, 94, 95, 106, 93, 96 | 0 | 0 | 2 | 1 | 1 | 0
  UP, 3+, BL, n=92, 94, 95, 106, 93, 96 | 1 | 1 | 0 | 0 | 0 | 0
  UP, Neg, BL, n=92, 94, 95, 106, 93, 96 | 70 | 76 | 80 | 89 | 80 | 78
  UP, Trace, BL, n=92, 94, 95, 106, 93, 96 | 14 | 10 | 7 | 8 | 7 | 14
  UP, 1+, W8, n=71, 81, 82, 93, 82, 77 | 3 | 2 | 5 | 1 | 4 | 2
  UP, 2+, W8, n=71, 81, 82, 93, 82, 77 | 2 | 1 | 0 | 1 | 1 | 0
  UP, 3+, W8, n=71, 81, 82, 93, 82, 77 | 0 | 0 | 0 | 0 | 1 | 0
  UP, Neg, W8,n=71, 81, 82, 93, 82, 77 | 60 | 70 | 68 | 78 | 64 | 71
  UP, Trace, W8, n=71, 81, 82, 93, 82, 77 | 6 | 8 | 9 | 13 | 12 | 4
  UP, Neg, EW, n=2, 1, 2, 3, 1, 7, 1, 7 | 2 | 1 | 2 | 3 | 1 | 5
  UP, Trace, EW, n=2, 1, 2, 3, 1, 7 | 0 | 0 | 0 | 0 | 0 | 2
  UWBC, 1+, BL, n=92, 94, 95, 106, 93, 96 | 1 | 1 | 6 | 1 | 6 | 3
  UWBC, 2+, BL, n=92, 94, 95, 106, 93, 96 | 1 | 3 | 1 | 7 | 2 | 3
  UWBC, 3+, BL, n=92, 94, 95, 106, 93, 96 | 0 | 3 | 2 | 2 | 1 | 2
  UWBC, Mod, BL, n=92, 94, 95, 106, 93, 96 | 0 | 0 | 0 | 0 | 1 | 0
  UWBC, Neg, BL, n=92, 94, 95, 106, 93, 96 | 88 | 84 | 82 | 92 | 81 | 85
  UWBC, Trace, BL, n=92, 94, 95, , 93, 96 | 2 | 3 | 4 | 4 | 2 | 3
  UWBC, 1+, W8, n=71, 81, 82, 93, 82, 77 | 1 | 3 | 2 | 3 | 7 | 4
  UWBC, 2+, W8, n=71, 81, 82, 93, 82, 77 | 1 | 1 | 4 | 3 | 2 | 3
  UWBC, 3+, W8, n=71, 81, 82, 93, 82, 77 | 0 | 0 | 2 | 1 | 0 | 1
  UWBC, Neg, W8, n=71, 81, 82, 93, 82, 77 | 66 | 71 | 69 | 81 | 67 | 67
  UWBC, Small, W8, n=71, 81, 82, 93, 82, 77 | 1 | 0 | 1 | 0 | 0 | 0
  UWBC, Trace, W8, n=71, 81, 82, 93, 82, 77 | 2 | 6 | 4 | 5 | 6 | 2
  UWBC, 2+, EW, n=2, 1, 2, 3, 1, 7 | 0 | 1 | 0 | 0 | 0 | 1
  UWBC, Neg, EW, n=2, 1, 2, 3, 1, 7 | 2 | 0 | 2 | 3 | 1 | 6

19. Secondary Outcome: Urine Specific Gravity at Baseline and Week 8/Early Withdrawal
Description: Urine samples were collected for the measurement of urine specific gravity by dipstick method at Baseline and at Week 8/Early Withdrawal. The Baseline value was the measurement taken at screening (Visit 1). Specific gravity is a measure of the amount of material dissolved in the urine. Specific gravity is the ratio of the density (mass of a unit volume) of a substance to the density (mass of the same unit volume) of a reference substance. Normal urine has a specific gravity between 1.010 and 1.020.
Time Frame: Baseline and Week 8/Early Withdrawal
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Placebo | GW685698X 25 µg OD | GW685698X 50 µg OD | GW685698X 100 µg OD | GW685698X 200 µg OD | FP 100 µg BID
Number analyzed (Participants) | 94 | 97 | 100 | 110 | 95 | 102
ratio
  Baseline, n=92, 94, 95, 106, 93, 96 | 1.0230 (0.00707) | 1.0240 (0.00690) | 1.0236 (0.00682) | 1.0230 (0.00687) | 1.0242 (0.00620) | 1.0227 (0.00760)
  Week 8, n=71, 81, 82, 93, 82, 77 | 1.0238 (0.00731) | 1.0227 (0.00735) | 1.0230 (0.00714) | 1.0223 (0.00738) | 1.0235 (0.00727) | 1.0217 (0.00751)
  EW, n=2, 1, 2, 3, 1, 7 | 1.0265 (0.00071) | 1.0121 (0) | 1.0200 (0.00141) | 1.0233 (0.00987) | 1.0190 (0) | 1.0240 (0.00653)

20. Secondary Outcome: Urine pH at Baseline and Week 8/Early Withdrawal
Description: Urine samples were collected for the measurement of urine pH by dipstick method at Baseline and at Week 8/Early Withdrawal. The Baseline value was the measurement taken at screening (Visit 1). Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acid pH (5.0 - 6.0).
Time Frame: Baseline and Week 8/Early Withdrawal
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | GW685698X 25 µg OD | GW685698X 50 µg OD | GW685698X 100 µg OD | GW685698X 200 µg OD | FP 100 µg BID
Number analyzed (Participants) | 94 | 97 | 100 | 110 | 95 | 102
scores on a scale
  Baseline, n=92, 94, 95, 106, 93, 96 | 6.04 (0.487) | 6.05 (0.418) | 6.06 (0.455) | 6.13 (0.488) | 6.05 (0.489) | 6.08 (0.415)
  Week 8, n=71, 81, 82, 93, 82, 77 | 6.03 (0.422) | 6.01 (0.418) | 6.12 (0.462) | 6.06 (0.435) | 6.06 (0.523) | 5.96 (0.342)
  EW, n=2, 1, 2, 3, 1, 7 | 6.00 (0.707) | 6.00 (0) | 5.75 (0.354) | 6.83 (0.289) | 7.50 (0) | 5.86 (0.556)

21. Secondary Outcome: 24-hour Urinary Cortisol Excretion at Baseline and Week 8
Description: A 24-hour urine sample was collected for the measurement of 24 hr urinary cortisol excretion at the following scheduled time points: within 7 days prior to Study Visits 3 (Week 0) and Visit 8 (Week 8). The Baseline value for 24 hr urinary cortisol was taken from Visit 3.
Time Frame: Baseline and Week 8
Population: Urine Cortisol (UC) Population: all participants whose urine samples did not have confounding factors that could affect the interpretation of results.
Measure: Median (Full Range); unit: Nanomoles per 24 hours (nmol/24 hours)
Arm/Group | Placebo | GW685698X 25 µg OD | GW685698X 50 µg OD | GW685698X 100 µg OD | GW685698X 200 µg OD | FP 100 µg BID
Number analyzed (Participants) | 66 | 72 | 72 | 76 | 69 | 70
Nanomoles per 24 hours (nmol/24 hours)
  Baseline | 70.20 [10.1 to 382.7] | 74.45 [6.1 to 645.2] | 65.80 [5.9 to 341.1] | 65.56 [8.8 to 457.3] | 66.80 [4.6 to 396.2] | 66.20 [6.4 to 338.6]
  Week 8 | 79.25 [7.5 to 275.0] | 76.74 [5.2 to 306.6] | 79.15 [13.9 to 680.9] | 81.0 [10.6 to 506.6] | 62.10 [8.0 to 366.7] | 82.14 [4.7 to 231.0]

22. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at Week 8
Description: Change from Baseline was calculated as the Week 8 value minus the Baseline value.
Time Frame: Baseline and Week 8
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Placebo | GW685698X 25 µg OD | GW685698X 50 µg OD | GW685698X 100 µg OD | GW685698X 200 µg OD | FP 100 µg BID
Number analyzed (Participants) | 78 | 85 | 91 | 98 | 86 | 84
Millimeters of mercury (mmHg)
  SBP | -2.5 (9.29) | 1.5 (10.54) | 0.9 (10.35) | -0.4 (10.46) | 1.4 (9.53) | 0.2 (10.64)
  DBP | -1.1 (8.16) | 0.3 (7.65) | 0.2 (7.50) | -0.3 (8.41) | 0.1 (8.50) | -0.2 (8.55)

23. Secondary Outcome: Change From Baseline in Heart Rate at Week 8
Description: Change from Baseline was calculated as the Week 8 value minus the Baseline value.
Time Frame: Baseline and Week 8
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | GW685698X 25 µg OD | GW685698X 50 µg OD | GW685698X 100 µg OD | GW685698X 200 µg OD | FP 100 µg BID
Number analyzed (Participants) | 78 | 85 | 91 | 98 | 86 | 84
Beats per minute | 2.9 (9.23) | 0.4 (8.26) | 1.5 (8.35) | 0.8 (8.12) | -2.3 (8.32) | 0.8 (9.14)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the start of study medication to the end of the the treatment period (up to Week 8).
Description: SAEs and non-serious AEs were reported for members of the Intent-to-Treat (ITT) Population, comprised of all participants randomized to treatment who received at least one dose of trial medication during the treatment period.
Arm/Group | Placebo | GW685698X 25 µg OD | GW685698X 50 µg OD | GW685698X 100 µg OD | GW685698X 200 µg OD | FP 100 µg BID
Serious Adverse Events (participants affected / at risk) | 0/94 | 1/97 | 0/100 | 1/110 | 0/95 | 2/102
Other Adverse Events (participants affected / at risk) | 11/94 | 6/97 | 8/100 | 17/110 | 9/95 | 16/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=94) | GW685698X 25 µg OD (N=97) | GW685698X 50 µg OD (N=100) | GW685698X 100 µg OD (N=110) | GW685698X 200 µg OD (N=95) | FP 100 µg BID (N=102)
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Snake bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=94) | GW685698X 25 µg OD (N=97) | GW685698X 50 µg OD (N=100) | GW685698X 100 µg OD (N=110) | GW685698X 200 µg OD (N=95) | FP 100 µg BID (N=102)
Headache (Nervous system disorders) | 10 | 6 | 6 | 12 | 5 | 12
Oropharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 4 | 3 | 2
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 4 | 3 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.